CLINICAL TRIAL: NCT02133118
Title: A Prospective Observational Cohort Study; The Weight Trajectory in New Users of Sulfonylureas as Add on Therapy Next to Metformin.
Brief Title: Weight Trajectory in New Users of Sulfonylureas as Add on Therapy Next to Metformin.
Acronym: ZODIAC-39
Status: Completed | Type: Observational
Sponsor: Medical Research Foundation, The Netherlands (Other)
Responsible Party: Principal Investigator, Gijs Landman, MD, PHD, Medical Research Foundation, The Netherlands
Other Study IDs: ZODIAC
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; New-user design; Weight trajectory; Add-on therapy; Sulphonylureas.
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Body-Weight Trajectory | interventions — Insulin; Pioglitazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients on metformin mono-therapy who receive add-on
  Interventions: Drug: individual SUs, insulin, pioglitazone

INTERVENTIONS:
Drug: individual SUs, insulin, pioglitazone

SUMMARY:
Next to HbA1c, body weight is regarded as an important surrogate end-point in trials investigating glucose-lowering agents. An increase in weight could contribute to worsening insulin resistance. Differences in weight after starting glucose lowering agents have been described in many randomized controlled trials (RCTs).

With this prospective observational study, weight trajectories after receiving add-on therapy next to metformin are evaluated in primary care patients with good glycaemic control.

DETAILED DESCRIPTION:
This prospective cohort study is part of the ZODIAC (Zwolle Outpatient Diabetes project Integrating Available Care) study, which started in 1998 as a prospective observational study and includes patients with known T2DM who are treated in primary care.

The investigators aim to investigate the course of the bodyweight and glycaemic control, the years after starting specific SU's, pioglitazone or insulin as add-on therapy, in metformin treated primary care patients with T2DM.

As part of the process called benchmarking, a dataset of quality measures is collected annually for all patients participating in the ZODIAC study during the patient's visit to the practice nurse and/or general practitioner and sent to the investigators' diabetes centre for benchmarking and research purposes once a year.

ELIGIBILITY:
Inclusion Criteria:

* T2DM
* Treated in primary care in period 1998 to 2012
* used metformin monotherapy
* subsequently received add-on therapy with a SU or pioglitazone during their entire follow-up period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with T2DM who received monotherapy with metformin and needed treatment intensification by receiving add-on therapy next to metformin
Sampling Method: Non-Probability Sample
Enrollment: 16293 (Actual)
Dates: Start 1998-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The course of weight (Kg) after starting individual SU's, pioglitazone or insulin as add-on therapy. | Up to 5 years
  The course of the bodyweight up to five years after starting individual SU's (gliclazide/glibenclamide/tolbutamide/glimepiride), pioglitazone or insulin as add-on therapy, in metformin treated primary care patients with T2DM.

SECONDARY OUTCOMES:
The course of the glycaemic control (HbA1c %) , up to five years after starting individual SU's, pioglitazone or insulin as add-on therapy. | Up to 5 years
  The course of the glycaemic control, up to five years after starting individual SU's (gliclazide, glibenclamide, tolbutamide, glimepiride), pioglitazone or insulin as add-on therapy, in metformin treated primary care patients with T2DM.

CONTACTS AND LOCATIONS:
Overall Officials: G. W.D. Landman, MD PhD, Principal Investigator — Isala, Diabetes Centre; R. Wever, MD, Principal Investigator — Isala, Diabetes Centre; P. R. van Dijk, MD, Principal Investigator — Isala, Diabetes Centre; Nanne Kleefstra, MD PhD, Study Director — Diabetes Centre, Isala, Zwolle
Locations (1):
- Isala, Zwolle, Overijssel, Netherlands